CLINICAL TRIAL: NCT04728438
Title: Effect of Targeted Temperature Management on Cerebral Autoregulation in Patients With Neurocritical Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202101005
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-12

CONDITIONS: Ischemic Stroke; Subarachnoid Hemorrhage, Aneurysmal; Sepsis; TBI (Traumatic Brain Injury); ICH - Intracerebral Hemorrhage; HIE - Hypoxic - Ischemic Encephalopathy
Keywords: cerebral autoregulation, targeted temperature management
MeSH Terms: conditions — Ischemic Stroke; Subarachnoid Hemorrhage; Sepsis; Brain Injuries, Traumatic; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Change and effect of cerebral autoregulation during targeted temperature management in neurocritical patients

DETAILED DESCRIPTION:
Cerebral autoregulation (CA) is the ability of cerebral vascular system to contract or diastole with the change of perfusion pressure, and to maintain the stability of cerebral blood flow. It has been found that there are different degrees of CA damage in patients with traumatic brain injury, ischemic stroke, hemorrhagic stroke, aneurysmal subarachnoid hemorrhage, ischemic hypoxic encephalopathy and sepsis. At the same time, studies have shown that CA damage or loss is related to brain dysfunction and poor prognosis in patients with neurocritical diseases. Therefore, early assessment and intervention of CA can help identify individuals with high risk of complications and improve outcome.

Targeted temperature management (TTM) is a kind of body temperature management started when the core temperature of patients is higher than 37.5 ℃, including achieve hypothermia (TTMhypo) and maintain normal temperature (TTMnorm). TTMhypo has been widely considered as one of the neuroprotective therapies for a variety of brain diseases and injuries, including ischemic stroke, traumatic brain injury, hypoxic brain injury caused by out-of-hospital cardiac arrest and neonatal hypoxic ischemic encephalopathy. Its neuroprotective effects in reducing brain edema, reducing intracranial pressure, reducing brain metabolism and inhibiting apoptosis have been recognized. However, the existing studies mainly focus on the effect of TTMhypo on the mortality and neurological outcome of patients with severe neurological diseases in ICU. There is no large clinical study on the effect of targeted temperature management (TTM) on cerebral autoregulation in patients with severe neurological diseases. Due to the controversy of TTMhypo on mortality and neurological outcome, this study aime to reduce the patient's core temperature to normal. Patients with severe neurological disorders who still had cerebral autoregulation dysfunction, had fever, and needed to reduce the core temperature to normal. Therefore, the effect of TTMnorm on cerebral autoregulation before and during cooling was observed.The main measures were the THRR, Mx and TOx during cooling.

ELIGIBILITY:
Inclusion Criteria:

- Aneurysmal subarachnoid hemorrhage (aSAH), Traumatic brain injury (TBI), Acute ischemic stroke (AIS), Intracerebral hemorrhage (ICH), Ischemic hypoxic encephalopathy (HIE), sepsis-associated encephalopathy (SAE) who need to reduce the core temperature to normal.

Exclusion Criteria:

* Age < 18 years old;
* Pregnancy;
* The temporal window was limited and the image could not be obtained;
* Patients with bradycardia induced by common carotid artery compression and intolerant of THRT
* Patients with severe carotid artery disease;
* Uncorrected severe coagulation disorders and active bleeding;
* Patients without informed consent;
* Patients who had been treated with hypothermia before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who need to reduce the core temperature to normal
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-22 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
discharge mortality | mortality when patients discharge，an average of 7days
  Mortality of patients included in the study

CONTACTS AND LOCATIONS:
Overall Officials: Lina Zhang, PhD, Study Chair — Xiangya University,Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China